CLINICAL TRIAL: NCT05137587
Title: Importance of Integrated Pulmonary Index in Pediatric Patients Undergoing Bronchoscopy Procedures Under Sedation
Brief Title: Importance of Integrated Pulmonary Index in Pediatric Bronchoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ruslan Abdullayev, Assist. Prof., Marmara University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 09.2021.497
Record Dates: First submitted 2021-11-25; First posted 2021-11-30 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2023-02

CONDITIONS: Monitored Anesthesia Care; Respiratory Monitoring
MeSH Terms: interventions — Propofol; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group P (Active Comparator): Patients sedated with propofol
  Interventions: Device: Integrated Pulmonary Index (IPI) monitoring; Drug: propofol
- Group K (Active Comparator): Patients sedated with ketamine
  Interventions: Device: Integrated Pulmonary Index (IPI) monitoring; Drug: ketamine

INTERVENTIONS:
Device: Integrated Pulmonary Index (IPI) monitoring — Integrated Pulmonary Index (IPI) monitor will be applied to the patients, to provide numerical data obtained from the measurements of end-tidal carbon dioxide, respiratory rate, oxygen saturation measured by pulse oximetry (SpO2), and pulse rate.
Drug: propofol — propofol
  Arms: Group P
Drug: ketamine — ketamine
  Arms: Group K

SUMMARY:
Integrated Pulmonary Index (IPI) is a tool that provides numerical values on a scale of 1-10 based on physiological parameters such as peripheral oxygen saturation (SpO2), pulse rate, respiratory rate, end-tidal carbon dioxide (ETCO2). It is a valuable monitor for sedation procedures and can provide early warning during cardiorespiratory derangements. In this study, we wanted to evaluate the value of IPI in cases of pediatric bronchoscopy performed under sedation. Our outcome measure will be the correlation of IPI values with standard monitoring parameters.

DETAILED DESCRIPTION:
Bronchoscopy is a procedure that is frequently applied in diagnostic or interventional conditions like hemoptysis, tracheobronchial stenosis, malignancy, recurrent lung infections, etc. It is routinely performed under general anesthesia or sedation in pediatric cases. In our clinic, we routinely perform diagnostic or interventional pediatric bronchoscopy procedures with an anesthesia team outside the operating room under monitored anesthetic care (MAC). Routine monitoring of MAC consists of electrocardiography (ECG), non-invasive blood pressure (NIBP), and peripheral oxygen saturation (SpO2). These monitorizations are described as minimum in many practice guidelines, and sometimes monitors such as end-tidal carbon dioxide (ETCO2), body temperature, analgesia/nociception index (ANI) can be added to them.

Integrated Pulmonary Index (IPI) is a tool that provides numerical values on a scale of 1-10 based on physiological parameters such as peripheral oxygen saturation (SpO2), pulse rate, respiratory rate, end-tidal carbon dioxide (ETCO2).(1,2) When these parameters exceed physiological limits, patients require interventions consisting of various maneuvers or drug administration in order to maintain the normal functioning of the cardiorespiratory system. If we look at the scoring, a score of 8-10 is considered normal, a score of 5-7 indicates a situation that may require intervention, and a score of 1-4 indicates that the patient needs intervention.

The above-mentioned IPI is a relatively new tool, and there is limited data in the literature regarding its usability in patients undergoing interventional procedures under MAC.(3,4) In this study, we wanted to evaluate the safety of IPI in cases of pediatric bronchoscopy performed under sedation. Routine monitoring and drug applications for the procedure will be in accordance with the institutional protocols, and additional IPI monitoring will be performed. Our outcome measure will be the correlation of IPI values with standard monitoring parameters.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3 physical status
* Elective upper or lower gastrointestinal tract endoscopy

Exclusion Criteria:

* ASA physical status of 4 or more
* Patients with any contraindication for off-site anesthesia

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
IPI-Ketamine | Throughout the sedation procedure
  Correlation of ketamine and IPI values

CONTACTS AND LOCATIONS:
Overall Officials: Ruslan Abdullayev, Principal Investigator — Marmara University Department of Anesthesiology and Reanimation
Locations (1):
- Marmara University School of Medicine, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taft A, Ronen M, Epps C, Waugh J, Wales R. A Novel Integrated Pulmonary Index (IPI) quantifies heart rate, etCO2, respiratory rate and SpO2%. ASA A1682, 22 Oct 2008.
- [Background] Berkenstadt H, Ben-Menachem E, Herman A, Dach R. An evaluation of the Integrated Pulmonary Index (IPI) for the detection of respiratory events in sedated patients undergoing colonoscopy. J Clin Monit Comput. 2012 Jun;26(3):177-81. doi: 10.1007/s10877-012-9357-x. Epub 2012 Mar 28. PMID 22454276
- [Background] Riphaus A, Wehrmann T, Kronshage T, Geist C, Pox CP, Heringlake S, Schmiegel W, Beitz A, Meining A, Muller M, von Delius S. Clinical value of the Integrated Pulmonary Index(R) during sedation for interventional upper GI-endoscopy: A randomized, prospective tri-center study. Dig Liver Dis. 2017 Jan;49(1):45-49. doi: 10.1016/j.dld.2016.08.124. Epub 2016 Sep 1. PMID 27671621
- [Background] Garah J, Adiv OE, Rosen I, Shaoul R. The value of Integrated Pulmonary Index (IPI) monitoring during endoscopies in children. J Clin Monit Comput. 2015 Dec;29(6):773-8. doi: 10.1007/s10877-015-9665-z. Epub 2015 Feb 11. PMID 25666393